CLINICAL TRIAL: NCT01305655
Title: Glucarpidase (CPG2) Effect on Severe Delayed Methotrexate-clearance in Children Treated With High-dose Methotrexate in Acute Lymphoblastic Leukemia (ALL)
Brief Title: Glucarpidase Effect on Severe Delayed HDM-clearance in Children Treated With High-dose Mtx in ALL
Acronym: NOPHOCPG2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Society for Pediatric Hematology and Oncology (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Heldrup, MD, Nordic Society for Pediatric Hematology and Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO2008CPG2
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: Drug: Glucarpidase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — glucarpidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucarpidase arm (Experimental): In the NOPHO ALL-2008 protocol patients with delayed methotrexate elimination (DME) in high-dose methotrexate treatments should be given Glucarpidase (50 ie/kg) with-in 60 hours from start of the methotrexate treatment.
  Interventions: Drug: Glucarpidase

INTERVENTIONS:
Drug: Glucarpidase — Patients treated with Glucarpidase if the 24 hour levels of MTX is >250 µM, 36 hour levels >30 µM or 42 hours levels >10 µM together with a reduced kidney function will be compared with patients in just below the tricking values.
  Other Names: VORAXAZE®

SUMMARY:
Early intervention in children and adolescents who experience delayed MTX-clearance and renal dysfunction in ALL treatments with the enzyme Glucarpidase which rapidly hydrolyses MTX to non-toxic metabolites to avoid life threatening complications.

DETAILED DESCRIPTION:
The NOPHO ALL-2008 protocol is a treatment and research protocol that aims to improve the overall outcome of Nordic children and adolescents with ALL in comparison with the ALL-2000 protocol and with the aim to reduce and prevent toxic treatment complications with high-dose methotrexate (HD-MTX).

The specific and primary objectives of the randomized study is:

1. Early intervention in children and adolescents who experience delayed MTX-clearance and renal dysfunction with the enzyme Glucarpidase which rapidly hydrolyses MTX to non-toxic metabolites and lowers the serum concentration to avoid life threatening complications. Glucarpidase should be given if the 24 hour levels of MTX is > 250 µM, 36 hour levels > 30 µM or 42 hours levels > 10 µM together with a reduced kidney function. Glucarpidase treatment should take place within 48 hours from the start of HD-MTX treatment.
2. To evaluate if the early intervention with Glucarpidase reduce the number of days the patients have to stay at the hospital.
3. Evaluate the reduction of health costs of early intervention in patients with delayed MTX-clearance and renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents who experience delayed MTX-clearance and renal dysfunction during high-dose methotrexate treatment in NOPHO ALL-2008.

Exclusion Criteria:

Children and adolescents with earlier anaphylactic reaction to Glucarpidase. Pregnant patients.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2008-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Heldrup, M D, Principal Investigator — University Childrens hospital, Lund, Sweden
Locations (5):
- Department of Pediatrics, Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- University of Reykjavik, Reykjavik, Iceland
- University Hospital of Trondheim, Trondheim, Norway
- Department of Pediatrics, Drottning Sylvias Pediatric Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Publication in preparation in Pediatric Blood and Cancer

REFERENCES:
- [Derived] Svahn T, Mellgren K, Harila-Saari A, Asberg A, Kanerva J, Jonsson O, Vaitkeviciene G, Stamm Mikkelssen T, Schmiegelow K, Heldrup J. Delayed elimination of high-dose methotrexate and use of carboxypeptidase G2 in pediatric patients during treatment for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2017 Jul;64(7). doi: 10.1002/pbc.26395. Epub 2016 Dec 14. PMID 27966809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 children treated with the NOPHO ALL 2008 protocol (1-18 years) in the Nordic- and Baltic countries received Glucarpidase if they had delayed Mtx elimination in connection HDMTX 5 g/sqr at predefined values.
Groups:
- Glucarpidase Arm: In children treated with high dose MTX (HDMTX) according to the NOPHO ALL 2008 protocol, Glucarpidase was used in case of predefined toxic MTX values at defined time points in combination with decreased renal function.
Period: Overall Study
Arm/Group | Glucarpidase Arm
Started | 47 (July 2008)
Completed | 47 (December 31, 2014)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glucarpidase Arm
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] — Children 1-18 years
  years | 7.5 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Region of Enrollment [Number; unit: participants]
  Sweden | 14
  Norway | 16
  Finland | 1
  Denmark | 11
  Iceland | 2
  Lithuania | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event to HD-MTX Treatment in NOPHO ALL-2008 as a Measure of Toxic Mtx Concentrations in Blood, Nephrotoxicity, Hepatotoxicity, Mucositis, MTX Elimination Time and Permanent Kidney Damage.
Description: Glucarpidase was used in case of predefined toxic MTX values at defined time points and/or in combination with decreased renal function.
  A total of 47 patients of the 1286 ALL-patients included in the protocol (3.7 %) were treated with Glucarpidase.
Time Frame: 6 years 6 months
Measure: Number; unit: participants
Groups:
- Glucarpidase Arm: 47 children treated with high dose MTX (HDMTX) according to the NOPHO ALL 2008 protocol, Glucarpidase was used in case of predefined toxic MTX values at defined time points in combination with decreased renal function.
Arm/Group | Glucarpidase Arm
Number analyzed (Participants) | 47
participants | 47

ADVERSE EVENTS:
Time Frame: 6 year, 6 months
Description: Non
Groups:
- Glucarpidase Arm: In the NOPHO ALL-2008 protocol patients with delayed methotrexate elimination (DME) in high-dose methotrexate treatments should be given Glucarpidase (50 ie/kg) with-in 60 hours from start of the methotrexate treatment.
  Glucarpidase: Patients treated with Glucarpidase if the 24 hour levels of MTX is >250 µM, 36 hour levels >30 µM or 42 hours levels >10 µM together with a reduced kidney function will be compared with patients in just below the tricking values.
  No serious effect reported.
Arm/Group | Glucarpidase Arm
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes